CLINICAL TRIAL: NCT05273268
Title: ZOE METHOD Study: Measuring Efficacy THrough Outcomes of Diet
Brief Title: ZOE METHOD Study: Comparing Personalized vs. Generalized Nutrition Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoe Global Limited (Other)
Collaborators: Massachusetts General Hospital (Other); Stanford University (Other); Harvard School of Public Health (HSPH) (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ZOE METHOD Study
Record Dates: First submitted 2022-02-18; First posted 2022-03-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Personalized Nutrition
Keywords: Gut microbiome; Personalized nutrition; Machine learning; Postprandial metabolism; Metabolic health

STUDY DESIGN:
Intervention Model Description: A randomised control trial with two parallel arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Active Comparator): The control arm (target enrollment; n=180) will receive the US government-standard guidelines for dietary advice in the form of the USDA dietary recommendations digital leaflet.
  Interventions: Other: Generalized nutrition
- Intervention Arm (Experimental): The intervention arm (target enrollment; n=180) will receive personalized dietary guidelines created by machine learning algorithms using their personal anthropometric, gut, dietary and medical information as inputs. The guidelines will be delivered in the form of a smartphone/ smart device app.
  Interventions: Other: Personalized nutrition

INTERVENTIONS:
Other: Personalized nutrition — Personalized nutrition based on individual traits delivered through mobile device app.
  Arms: Intervention Arm
Other: Generalized nutrition — General nutrition guidelines currently used by USDA.
  Arms: Control Arm

SUMMARY:
The ZOE Method Study will test the efficacy of personalized nutritional advice, delivered on an individual level through a digital device app; integrating dietary, lifestyle, physiological and metagenomic data, in improving certain cardiometabolic disease risk factors, compared to generalized nutrition advice (control).

DETAILED DESCRIPTION:
Personalized nutrition strategies offer potential for targeted dietary treatment and prevention of diet-related disease, and may ultimately serve as a powerful basis for stratified nutrition approaches at public health level. Existing research into personalized nutrition interventions has shown that it is superior compared to general advice when it comes to improving dietary quality, dietary behaviour, and dietary disease-risk biomarkers in a patient population with prediabetes. However, to date, the superiority of a personalized approach in improving the cardiometabolic risk phenotype in an apparently healthy adult population has not been investigated. With diet being an important modifiable factor for cardiometabolic disease risk, its preventative potential at a healthy individual level must be tested.

Public health policies aiming at reducing disease risk are traditionally derived from large-scale, low-precision epidemiological data that focuses on group means, leading to a 'one-size-fits-all' approach to nutritional guidelines. However, recent research shows that metabolic responses to foods and diet show huge variability at fasting and postprandially both within and between individuals, variation that is driven by 'what' we eat, 'how' we eat and 'who' we are. Metabolic responses to repeated dietary challenges are important underlying factors of diet-related disease risk. This warrants the integration of multiple dietary, lifestyle, physiological and metagenomic exposures into prescribed nutritional guidelines for effective disease risk prevention.

The ZOE METHOD Study will test the efficacy of such a personalized approach to nutritional guidance in improving cardiometabolic risk markers in a disease-free adult US population reflective of the general US phenotype.

Using a parallel randomized at-home design, this study will compare the effect of general dietary advice (USDA Dietary Guidelines for Americans) with the ZOE personalized dietary advice integrating exposures of 'what' we eat (logged free-living diet), 'how' we eat (lifestyle, meal context, time of day, exercise, sleep) and 'who' we are (physiological status and metagenomic signatures).

Population:

US adult subjects will be invited to take part in a 4-month long intervention with optional follow-ups at 8-12 months. A total of 360 participants will be enrolled onto the study with the aim of 300 participants completing the protocol (allowing for a drop-out rate of 20% given the remote nature of the study). Participants will be generally healthy, fall above the 25th percentile sex- and ethnicity-specific waist circumference (self-reported), and have fruit and vegetable intake below the 75th percentile of the US population (NHANES data). Participants will not have existing strict dietary patterns and will not be pregnant or breastfeeding, or not taking any medications that can alter glucose or lipid metabolism. Participants must also not be existing users of the product and must not have participated in any PREDICT studies to date.

Design:

The ZOE METHOD Study will take place remotely, with all study materials shipped to participants, in addition to 4 clinic-based blood draws at Quest Patient Centers. The study is marked by 4 timepoints (two at baseline, one mid-intervention, and one end-point) followed by two optional scheduled follow-ups.

Baseline 1:

Participant will complete two baselines; the first baseline (Week -1) consists of a visit to a Quest clinic to provide a fasted blood draw, blood pressure (BP), and anthropometric measurements (waist and hip circumference, body weight) while food frequency, lifestyle and health/medical history questionnaires are completed at home. BP and anthropometric measurements are also self-reported by the participant at home. Participants who do not complete their first Quest clinic visit will be withdrawn; those who successfully complete the first baseline are randomized to the control or intervention arm.

Randomization:

Participants will be assigned to either the intervention (ZOE personalized dietary advice) or control arm (USDA generalized dietary advice) once they have successfully completed Baseline 1 tasks.

Baseline 2:

The second baseline takes place one week after the first (Week 0) and consists of a second visit to a Quest clinic to provide anthropometry, BP and a fasted blood draw, followed by another questionnaire and at-home stool sample collection (for microbiome assessment). Both arms complete BP and anthropometric measurements at home again, as well as a fasted finger-prick dried blood spot test.

Treatment according to arm allocation starts at this second baseline; control participants are emailed a copy of the USDA Dietary Guidelines for Americans leaflet along with a short video where the dietary advice is explained. They are asked to follow this guidance.

Intervention participants receive the ZOE PREDICT 3 test kit, which they are asked to complete (thus partaking in multiple postprandial test meal challenges, providing continuous glucose measurements over 7-14 days, a postprandial triglyceride assessment by dried blood spot collection, and logged dietary intake) along with personalized ZOE dietary guidance.

Personalized dietary advice (Week 6 to Week 18):

Once their personalized nutritional guidance has been generated from the information collected in the testing phase (Week 0-2), the intervention group receives this personalized advice through a smart device. They are asked to complete a weighed food diary for 4 days after receiving their personalized dietary recommendations.

Both the control and intervention groups complete a health and lifestyle questionnaire at week 6. The control group continues following the USDA leaflet advice.

Mid-intervention measures (Week 12):

All participants complete a third Quest clinic visit to provide a fasted blood sample, BP and anthropometric measurements, as well as measuring these at home again alongside completing questionnaires and a stool sample collection. The intervention group is asked to complete a 4-day weighed food diary again at this time.

Endpoint measures (Week 18):

Both control and intervention participants complete their fourth Quest clinic assessment for anthropometry, BP and fasted blood collection, answer online questionnaires and provide a post-treatment stool sample, as well as completing a fasted finger-prick dried blood spot test, BP and anthropometric measures at home. The intervention group completes the ZOE test kit for the second time to assess postprandial triglyceride response and continuous glucose measurements, as well as a 4-day weighed food diary.

At this endpoint, control-group participants are given the option to complete the ZOE test kit and PREDICT 3. Control participants are also given the option of joining a nested cross-over arm following their 18 week Endpoint completion. Nested cross-over participants are asked to complete the intervention arm protocol, thus following the personalized dietary guidance received from the ZOE PREDICT 3 test kit and complete the Week 6, Week 12 and Week 18 checkpoints as required for intervention participants (thus including weighed food diaries).

Follow-ups:

Intervention participants are followed-up at Month 8 and again at Month 12 with a clinical visit, questionnaires, stool sample collection and at-home biometric measures.

Outcomes:

The ZOE METHOD Study will investigate the effect of following personalized approach to nutritional guidance vs. general nutritional guidelines on certain cardiometabolic and diet-related disease risk factors. The primary outcomes are low-density-lipoprotein cholesterol (LDL-C) and triglycerides (mmol/L) assessed at each fasted blood-draw. Secondary and exploratory outcomes are listed below, and include weight, waist circumference, BP, glycemic control, gut microbiome assessment, and self-reported hunger.

Assessment of postprandial metabolic responses :

Participants in the Intervention will be provided with a standardized dietary intervention in the form of muffins, to be consumed at breakfast on two days and a subsequent lunch meal on one day. Nested cross-over participants will receive one breakfast and one lunch meal to be consumed on one testing day. Participants are instructed to fast before and after these tests, but are free to eat and drink as they wish during the rest of the study. During this time participants will be wearing a continuous glucose monitor and will complete a 6 h finger-prick dried blood spot sample to assess triglycerides after their mixed sequential meal challenge (breakfast-lunch) test. This protocol is equivalent to that followed by PREDICT 3 participants (NCT04735835).

Participant Contact: Regular contact will be made with the participants via email, phone, their app and in-app messages for the period of the treatment to encourage compliance and answer any queries.

Health history, lifestyle and habitual intake information: Participants will be asked to complete multiple questionnaire online throughout the study, including the assessment of lifestyle aspects pertaining to nutrition (exercise, sleep) and eating habits and appetite, as well as health and medical history for the assessment of physiological status and potential genetic-derived risk scores, and finally their habitual dietary intake through a food-frequency questionnaire pertaining to the previous month with portion sizes. Intervention and nested cross-over participants will also be asked to log a weighed food diary using the ZOE app for up to 4 consecutive days per month (total of 4 logging periods), as well as a diet history questionnaire with portion sizes about the month preceding it's reporting (at Week 0, Week 12 and Week 18).

Outcome analysis may be stratified according to baseline combined fruit and vegetable intake, age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-70 years
* Any sex
* Waist circumference greater than ethnic- and sex-specific 25th percentile values:

Male

* Hispanic > 96.3cm
* Asian > 87.3cm
* Black > 92.7cm
* White > 96.9cm Female
* Hispanic > 90.7cm
* Asian > 80.9cm
* Black > 92.9cm
* White > 88.3cm

  * Fruit and vegetable intake below 450g/day (equivalent to 3 cups/day)
  * Willing to comply with study protocol
  * Live in the continental US, Hawaii or Alaska, and not in New York State (due to governmental regulations pertaining to dried blood spot testing).
  * Do not meet any of the exclusion criteria

Exclusion Criteria:

* Have taken part in the ZOE product or any PREDICT study beforehand.
* Are unable to read and write in English, as the ZOE app is only available in English.
* Do not complete the first Quest visit successfully
* Have an iOS/Android device not compatible with app
* Use medications affecting lipids (lipid lowering drugs e.g statins, anti-diabetic medications, e.g metformin and insulin), supplements including fish oil (unless willing to safely come off these for 4 weeks before the start of the study, and for the duration of study);
* Have ongoing inflammatory disease e.g rheumatoid arthritis, systemic lupus erythematosus, polymyalgia and other connective tissue diseases.
* Have had cancer in the last three years, excluding skin cancer.
* Have chronic gastrointestinal disorders including inflammatory bowel disease (IBD) or Celiac disease (gluten allergy), but not including irritable bowel syndrome (IBS).
* Are taking the following daily medications: immunosuppressants, corticosteroids, antibiotics in the last three months, not including inhalers.
* Are users of prescription proton pump inhibitors (PPIs) (such as omeprazole and pantoprazol), unless they are able to stop two weeks before the start of the study and remain off them for the entire duration of the study (provided their treating physician deems it safe for them to do so).
* Are currently suffering from acute clinically diagnosed depression or anxiety disorder.
* Have had a heart attack (myocardial infarction) or stroke in the last 6 months.
* Are pregnant or planning pregnancy in next 12 months, or are breastfeeding
* Are vegan, have an eating disorder or unwilling to take foods that are part of the study.
* Have an allergy to adhesives which would prevent proper attachment of the continuous glucose monitor.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Fasted blood lipids | 12 months (0 wk, 1 wk, 13 wk, 19 wk, 8mo, 12mo)
  Fasted measurement of triglycerides and LDL-cholesterol (mmol/L) by venous blood draw.

SECONDARY OUTCOMES:
Body weight | 12 months (0 wk, 1 wk, 7 wk, 13 wk, 19 wk, 8mo, 12mo)
  Body weight (kg)
Waist circumference | 12 months (0 wk, 1 wk, 7 wk, 13 wk, 19 wk, 8mo, 12mo)
  Waist circumference (cm)
Hip circumference | 12 months (0 wk, 1 wk, 7 wk, 13 wk, 19 wk, 8mo, 12mo)
  Hip circumference (cm).
Blood pressure | 12 months (0 wk, 1 wk, 7 wk, 13 wk, 19 wk, 8mo, 12mo)
  Measurement by clinical and home-based device (mmHg).
HbA1c | 12 months (0 wk, 19 wk, 8mo, 12mo)
  Fasted measurement by venous blood draw (%).
Insulin | 12 months (0 wk, 1 wk, 13 wk, 19 wk, 8mo, 12mo)
  Fasted measurement by venous blood draw (IU/L).
Glucose | 12 months (0 wk, 1 wk, 13 wk, 19 wk, 8mo, 12mo)
  Fasted measurement by venous blood draw (mmol/L).
C-peptide | 12 months (0 wk, 19 wk, 8mo, 12mo)
  Fasted measurement by venous blood draw (mmol/L).
Apo-B and Apo-A | 12 months (0 wk, 19 wk, 8mo, 12mo)
  Fasted measurement by venous blood draw (mmol/L).
Gut microbiome health | 12 months (0 wk, 1 wk, 13 wk, 19 wk, 8mo, 12mo)
  Gut microbiome assessment from stool sample for species richness and diversity.
Postprandial triglyceride level | 19 weeks (1 wk, 19 wk)
  Measured at 6 hours following a breakfast-lunch test meal challenge (intervention only; mmol/L).
Habitual diet quality | 12 months (1 wk, 13 wk, 19 wk, 8 mo, 12 mo)
  Self-reported habitual diet quality assessed by food frequency questionnaire.
Energy level | 12 months (1 wk, 7 wk, 13 wk, 19 wk, 8 mo, 12 mo)
  Self-reported energy level by questionnaire.

OTHER OUTCOMES:
Glycemic control (Intervention arm only) | 19 weeks (1 wk, 19 wk)
  Glucose time in range and postprandial continuous glucose quantification, derived from continuous glucose sensor used in Intervention Arm only.
hsCRP | 12 months (0 wk, 1 wk, 13 wk, 19 wk, 8mo, 12mo)
  hsCRP quantification in fasted venous blood draw (mmol/L).
Glycan markers | 19 weeks (1 wk, 19 wk)
  Glycan quantification in fasted dried blood spot tests.
Skin quality | 12 months (1 wk, 7 wk, 13 wk, 19 wk, 8 mo, 12 mo)
  Self-reported by questionnaire.
Mood | 12 months (1 wk, 7 wk, 13 wk, 19 wk, 8 mo, 12 mo)
  Self-reported by questionnaire.
Hunger | 12 months (1 wk, 7 wk, 13 wk, 19 wk, 8 mo, 12 mo)
  Self-reported by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Berry, PhD, Principal Investigator — King's College London and consultant at ZOE Ltd; Tim Spector, Pr, Principal Investigator — King's College London and consultant at ZOE Ltd
Locations (1):
- ZOE Ltd, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bermingham KM, Linenberg I, Polidori L, Asnicar F, Arre A, Wolf J, Badri F, Bernard H, Capdevila J, Bulsiewicz WJ, Gardner CD, Ordovas JM, Davies R, Hadjigeorgiou G, Hall WL, Delahanty LM, Valdes AM, Segata N, Spector TD, Berry SE. Effects of a personalized nutrition program on cardiometabolic health: a randomized controlled trial. Nat Med. 2024 Jul;30(7):1888-1897. doi: 10.1038/s41591-024-02951-6. Epub 2024 May 8. PMID 38714898